CLINICAL TRIAL: NCT04773405
Title: Minimum Effective Local Anaesthetic Volume of a 1:1 Mixture of 2% Lidocaine With 5ug/ml of Epinephrine and 0.5% Levobupivacaine Required for Ultrasound Guided Selective Trunk Block: A Dose Finding Study
Brief Title: Minimum Effective Volume for Selective Trunk Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SeTB MEV Ver 4
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Selective Trunk nerve block
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Lidocaine; Epinephrine; Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selective Trunk Block (Other): Selective trunk block will be done under ultrasound guidance to patients scheduled for upper extremities surgeries. Local anaesthetic agents (a 1:1 mixture of 2% lidocaine with 5ug/ml of epinephrine and 0.5% levobupivacaine) will be injected at the superior, middle, and inferior trunks of the brachial plexus in order to anaesthetize the whole upper limb.
  Interventions: Drug: a 1: 1 mixture of 2% lidocaine with 5ug/ml epinephrine and 0.5% levobupivacaine

INTERVENTIONS:
Drug: a 1: 1 mixture of 2% lidocaine with 5ug/ml epinephrine and 0.5% levobupivacaine — This study adopts a "Modified Narayana rule (MNR)", a sequential up-and-down pharmacodynamics method (UDM) to estimate the minimum effective local anesthetic volume of 90% (MELAV90) of cases of the aforementioned local anaesthetic (LA) mixture, in order to produce the surgical anaesthesia of the whole upper extremity of the patients scheduled for upper limb surgeries. Based on the principal investigator's clinical experience, the initial volume of 21ml will be used. Depending on the success or failure of the SeTB, which is defined as the readiness for surgery at 30 minutes after the block, the volume for the next patient will be adjusted up or down by 3ml (1ml for each trunk of brachial plexus located above the clavicle). The upper dose limit of the study to minimize the potential for local anaesthetic systemic toxicity will be 30ml and the lower dose limit will be 12ml, which will be of no clinical importance.
  Other Names: Selective trunk block

SUMMARY:
The objective of this study is to identify the minimum effective dosage of a mixture of two local anaesthetic drugs called 'levobupivacaine' and 'lignocaine with epinephrine" used to produce an effective ultrasound guided selective trunk block for surgical anaesthesia of the upper limb.

DETAILED DESCRIPTION:
Ultrasound is widely used for brachial plexus block (BPB) and current evidence indicates that it is feasible to accurately identify majority of the main components of the brachial plexus above the clavicle, including the three trunks. Since majority of the innervation to the upper extremity, including the shoulder, arises from the three trunks (superior, middle and inferior) of the brachial plexus, so targeted injections of the individual trunks of the brachial plexus under ultrasound guidance will produce surgical anaesthesia of the entire upper extremity (C5-T1). Principal Investigator refers to this novel technique "selective trunk block" (SeTB) and the preliminary experience with SeTB for surgical anaesthesia of the entire upper extremity has been very encouraging. Currently there are no data describing an optimal dose or volume of local anaesthetic for SeTB. The aim of this study is to identify the minimum dosage of 1:1 mixture of 'levobupivacaine' and "lignocaine with epinephrine" required to produce effective surgical anaesthesia in at least 90% of patients presented for upper limb surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III scheduled to undergo elective upper extremity surgery involving the proximal humerus to distal hand or surgery involving any combination of these regions.

Exclusion Criteria:

* Patient refusal
* pregnancy
* skin infection at the site of block placement
* history of allergy to local anaesthetic drugs
* history of bleeding tendency or with evidence of coagulopathy
* pre-existing neurological deficit
* pre-existing neuromuscular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Changes of sensory block of the upper extremity | within 45 minutes after the block at 5 minutes interval
  Sensation to coldness (ice) will be tested at C5 - Lateral (radial) side of the antecubital fossa (just proximal to elbow crease), C6 - Thumb, dorsal surface, proximal phalanx, C7 - middle finger, dorsal surface, proximal phalanx, C8 - Little finger, dorsal surface, proximal phalanx, and T1 - medial (ulnar) side of the antecubital) fossa, just proximal to the medial epicondyle of the humerus. Sensory block, defined as loss of sensation to cold (ice), will be graded using a numeric rating scale (NRS: 0-100, 100=normal sensation, 0=no sensation). A 3-point qualitative sensory score (0=no block, 1=analgesia/ patient can feel touch but not cold, and 2=anaesthesia / patient cannot feel touch) will be used. Onset of sensory block for each nerve will be defined as the time that it took to achieve a sensory block score of NRS =<30 and Qualitative sensory score =1 .
Changes of motor blockade of the upper extremity | within 45 minutes after the block at 5 minutes interval
  motor blockade will be graded using a 3-point scale: 0=no block, 1=paresis and 2=paralysis. Motor blockade of each individual nerve in the anaesthetized upper extremity will be evaluated by testing C5 - elbow flexors, C6 - Wrist extensors, C7 - Elbow extensors, C8 - Finger flexors to the middle finger, and T1 - small finger abductors. Onset of Motor block for each nerve will be defined as the time it took to achieve motor score >=1.
Readiness for surgery | within 45 minutes after the block at 5 minutes interval
  Overall sensory score of NRS =<30 (NRS: 0-100; 100=normal sensation, 0=no sensation) and Qualitative sensory score =1 for each nerve; and motor scores >=1 (3 point scale: 0=no block, 1=paresis, 2=paralysis) in all nerves tested. Overall the maximum composite sensory-motor score achievable is 20 points (2 points for each 5 sensory nerves tested and 2 points for each 5 motor nerves tested).

SECONDARY OUTCOMES:
Changes of the Diaphragmatic function | Baseline (before block) and at 30 minutes after block
  Excursion of the right hemidiaphragm will be measured by ultrasound machine in supine position via the anterior subcostal route. The movement of the diaphragm will be measured in centimetres. The range of diaphragmatic excursion will be recorded from the resting expiratory position to deep inspiration (sigh test) as will be the range of diaphragmatic movement from resting expiratory position when quickly inspiring through the nose (sniff test). The decrease in diaphragmatic excursion will be calculated as the difference (in %) in diaphragmatic excursion measured before and 30 minutes after SeTB. Reduction in diaphragmatic excursion of more than 75%, or no movement, or paradoxical movement will be considered as complete paresis. Reduction in diaphragmatic excursion of both sigh and sniff test between 25% and 75% will be considered as partial paresis and diaphragmatic excursion of less than 25% will be considered as 'no paresis'.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia & Intensive Care, Prince of Wales Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- [Derived] Sivakumar RK, Karmakar MK, Wong RSL, Samy W. Minimum effective volume 90% for ultrasound-guided selective trunk block: A quantal bioassay. Eur J Anaesthesiol. 2025 Sep 1;42(9):800-807. doi: 10.1097/EJA.0000000000002160. Epub 2025 Mar 11. PMID 40070288